CLINICAL TRIAL: NCT04667975
Title: A Multicenter, Open-Label, Dose-Escalation and Dose-Expansion, Phase I Study to Evaluate the Safety, Pharmacokinetics and Anti-tumor Effects of CKD-702 in Patients With Advanced or Metastatic Non-small Cell Lung Cancer Who Failed to Standard Therapy
Brief Title: The Purpose of Study is to Evaluate the Safety, Pharmacokinetics and Anti-tumor Effects of CKD-702 in Patients With Advanced or Metastatic Non-small Cell Lung Cancer Who Failed to Standard Therapy
Acronym: CKD-702
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 187NSCLC18021
Record Dates: First submitted 2020-09-29; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: * Part 1(Dose Escalation)
    1. Level 1(10mg/kg)
    2. Level 2(15mg/kg)
    3. Level 3(20mg/kg)
    4. Level 4(25mg/kg)
  * Part 2(Dose Expansion)
    1. EGFR TKI resistance
    2. EGFR Wild Type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1(Dose escalation) (Experimental): Part 1: 3 or 6 subjects are enrolled, per each dose group in a traditional 3+3 design.
  Begin with the starting dose determined by the non-clinical study and increase the dose according to the dose levels. If DLT does not occur in the 3 subjects when they have completed the 1st cycle at each dose level, increase the dose to the next level. Dose escalation proceeds until the maximum tolerated dose (MTD) is reached.
  Dose-limiting toxicity (DLT) is evaluated following the completion of dosing for the 1st cycle of all subjects enrolled in each dose group in order to determine whether to proceed to the next level. Following completion of the DLT evaluation of the planned dose level in this study, the SRC reviews the outcome of the evaluation and determines whether to set additional dosing or proceed to PART 2 (Dose expansion).
  Interventions: Drug: CKD-702
- Part 2(Dose expansion) (Experimental): Part 2: The primary objective of Part 2 is to evaluate the efficacy of CKD-702 by identifying the ORR after administering the RP2D of CKD-702 determined in Part 1. Along with this, to determine the CKD-702 effective patient group, the patient groups were classified into several cohorts based on non-clinical study results.
  Therefore, in Part 2, the RP2D determined in Part 1 is administered until the occurrence of an adverse event causing PD occurrence, death or treatment discontinuation, and tumor response is evaluated based on RECIST version 1.1.
  Interventions: Drug: CKD-702

INTERVENTIONS:
Drug: CKD-702 — In principle, based on 1 cycle of 28 days (4 weeks), administer CKD-702 Inj. once every 2 weeks over 4 weeks.

SUMMARY:
The purpose of study is to evaluate the safety, pharmacokinetics and anti-tumor effects of CKD-702 as a monotherapy and to determine the Recommended Phase 2 Dose(RP2D) in patients with advanced or metastatic non-small cell lung cancer who failed to standard therapy.

DETAILED DESCRIPTION:
This open label, multi center, first-in-human study consists of 2parts.

-Part 1: The dose is increased according to the prescribed dose escalation schedule.

Dose escalation proceeds until the maximum tolerated dose(MTD) is reached. Dose-limiting toxicity (DLT) is evaluated after completing cycle 1 administration for all subjects enrolled for each dose group in order to determine whether to proceed to the next level. all matters related to dose escalation are subject to the decision of the SRC. If DLT occurs in two subjects during the first dose level process, the dose level reset by the SRC is reflected and study protocol amendment procedure is followed accordingly. Following completion of the DLT evaluation of the planned dose level in this study, the SRC reviews the outcome of the evaluation and determines whether to set additional dosing or proceed to PART 2 (Dose expansion).

-Part 2: In Part 2, the recommended phase 2 dose (RP2D) of the CKD-702 Inj. determined in Part 1 is set as the treatment dose, and the dose must be administered with the same administration methods as Part 1, repeating cycles.

ELIGIBILITY:
Inclusion Criteria

1. Those aged 19 years or older
2. Patients with a definitive histological or cytological diagnosis of advanced or metastatic non-small-cell lung cancer (NSCLC) (according to the Cancer Staging Manual, AJCC/UICC, 8th ed., IIIB, IIIC and IV) and those for whom there was no applicable standard therapy or the standard therapy failed.
3. Those whose ECOG performance status is either 0 or 1
4. Patients who voluntarily decide to participate in this study and provide their written consent.

Exclusion Criteria

1. Patients whose toxicity due to previous anticancer therapy has not been reduced to Grade 1 or lower (However, hair loss of not less than Grade 2 and the peripheral neuropathy of Grade 2 are allowed)
2. Patients with malignant tumors other than NSCLC within the past 3 years of screening (However, treated local basal cell carcinoma or squamous cell carcinoma of skin, carcinoma in situ of uterine cervix, superficial bladder cancer, papillary thyroid carcinoma or, in the opinion of the investigator, malicious tumors that are considered to have little or no recurrence risk within 1 year, are permitted)
3. Patients with a history of serious heart disease such as acute ischemic heart disease within the past 6 months of screening (myocardial infarction, unstable angina, etc.) or heart failure of NYHA Class III or IV
4. Patients who have tested positive for HIV antibodies
5. Uncontrolled hypertension, diabetes patients
6. Patients who have not fully recovered from a major surgery or severe trauma before beginning treatment, or who are expected to undergo a major surgery during the study period or within 6 months of the final dose of the study drug.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose and/or Recommended Phase 2 Dose | Through study completion, an average of 2years
  To determine the maximum tolerated dose (MTD) and/or the recommended phase 2dose (RP2D)
Part 2: Objective Response Rate | Through study completion, an average of 2years
  To evaluate the objective response rate(ORR)

SECONDARY OUTCOMES:
Part 1(Dose Escalation): Pharmacokinetics(AUClast of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  1) AUClast of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics( AUCinf of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  2) AUCinf of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(Cmax of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  3) Cmax of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(t1/2 of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  4) t1/2 of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(Tmax of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  5) Tmax of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(CL of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  6) CL of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(Vz of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  7) Vz of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(MRT of CKD-702 after a single dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  8) MRT of CKD-702 after a single dose
Part 1(Dose Escalation): Pharmacokinetics(AUClast CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  9) AUClast CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(Cmax,ss CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  10) Cmax,ss CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(Cmin,ss CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  11) Cmin,ss CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(Cav,τ CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  12) Cav,τ CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(t1/2 CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  13) t1/2 CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(Tmax,ss CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  14) Tmax,ss CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(CLss CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  15) CLss CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(Vss CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  16) Vss CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(MRT CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  17) MRT CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(accumulation ratio CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  18) accumulation ratio CKD-702 after a repeated dose
Part 1(Dose Escalation): Pharmacokinetics(PTF of CKD-702 CKD-702 after a repeated dose) | C1D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs, C2D1 Pre-dose, Start of Infusion 0.5, 1hr, End of Infusion and End of Infusion 2, 6, 22, 70, 166, 336hrs
  19) PTF of CKD-702 CKD-702 after a repeated dose
Part 1(Dose Escalation): Immunogenicity(Analyze the idiotype antibody for hu8C4 (anti-cMET) Fab) | C1D1 Pre-dose, C1D15 Pre-dose, C2D1 Pre-dose, C3D1 Pre-dose, C4D1 Pre-dose,
  -Analyze the idiotype antibody for hu8C4 (anti-cMET) Fab
Part 1(Dose Escalation): Immunogenicity(Analyze the idiotype antibody for Vectibix scFv (anti-EGFR) | C1D1 Pre-dose, C1D15 Pre-dose, C2D1 Pre-dose, C3D1 Pre-dose, C4D1 Pre-dose,
  -Analyze the idiotype antibody for Vectibix scFv (anti-EGFR)
Part 2(Dose Expansion): Overall Survival | Through study completion, an average of 3years
  To evaluate overall survival (OS)
Part 2(Dose Expansion): Progression-Free Survival | Through study completion, an average of 3years
  To evaluate progression-free survival (PFS)
Part 2(Dose Expansion): Duration of Response | Through study completion, an average of 3years
  To evaluate the duration of response (DoR)
Part 2(Dose Expansion): Disease Control Rate | Through study completion, an average of 3years
  To evaluate the disease control rate (DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wan Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea